CLINICAL TRIAL: NCT03319979
Title: DHFR 19 bp Deletion Polymorphism and Folic Acid Utilization
Status: Completed | Type: Observational
Sponsor: Tufts University (Other)
Responsible Party: Sponsor
Other Study IDs: ORA# 1211023
Record Dates: First submitted 2017-10-20; First posted 2017-10-24 (Actual); Last update posted 2017-10-24 (Actual); Status verified 2017-10

CONDITIONS: Characterize rs70991108 Polymorphism of DHFR Gene
Keywords: Folate, DHFR

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
A genetic variation in the gene for the protein dihydrofolate reductase (DHFR) that is necessary to utilize folic acid (a synthetic form of the B vitamin folate found in supplements and fortified food), increases the risk for breast cancer in multivitamin users and, when present in mothers who used folic acid supplements during pregnancy, increases the risk for cancer of the eye of their children. The aim of the proposed research is to understand how a common genetic variation in the gene for DHFR affects the function of this protein and the ability of the body to use folic acid.

DETAILED DESCRIPTION:
A 19bp deletion polymorphism of intron 1 of dihydrofolate reductase (DHFR 19bpdel) increases the risk for breast cancer, and retinoblastoma of the offspring, in folic acid supplement users. Folic acid is a synthetic form of folate present in fortified foods and supplements that must be converted to tetrahydrofolate by DHFR to enter the metabolism. Individuals homozygous for DHFR 19bpdel have higher prevalence of unmetabolized folic acid in plasma and lower incorporation of folic acid into tissues. How the DHFR19bpdel (17% homozygosity in US) affects DHFR activity and folate metabolism to increase cancer risk is not understood. Studies on this topic are urgent in the light of mandatory folic acid fortification in the US and other countries. The objective of this project is to characterize the effect of DHFR 19bpdel on DHFR activity and folate pathway reactions and to determine if the effect of DHFR 19bpdel can be alleviated with folinic acid, which is a folate source that need not be converted by DHFR. The specific aims of this project are to 1] Determine expression of DHFR mRNA and protein, splicing of intron 1 and enzyme activity in white blood cells from 3 DHFR genotypes. 2] Determine the effect of DHFR 19bpdel and folic acid or folinic acid concentration on cell growth, and folate pathway reactions in white blood cells in homozygotes for DHFR 19bpdel and those who lack the polymorphism. Results of this study will guide measures to reduce this modifiable cancer risk associated with DHFR 19bpdel.

ELIGIBILITY:
Inclusion Criteria:

* Adult premenopausal women aged 21-45 in general good health, non-pregnant, minimum weight of 110 pounds.

Exclusion Criteria:

* Smoking, a terminal illness, any known chronic illness, rheumatoid arthritis, heart, kidney, liver or gastrointestinal disease requiring treatment, antifolate medications, metformin use.
* More than 2 drinks a day.
* Pregnant women have different metabolism when compared to other adults hence they will not be included in the study.
* Non-English speaking subjects will be excluded since the study involves a computer based diet history questionnaire in English. The budget for this project does not include the cost of an interpreter.

Ages: 21 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pre-menopausal women
Study Population: Healthy pre-menopausal females aged 21-45 from Metro Boston area
Sampling Method: Probability Sample
Enrollment: 117 (Actual)
Dates: Start 2013-02; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
DHFR mRNA and protein abundance | 1 year
  DHFR mRNA and protein abundance determined for the 19 bp deletion genotypes

SECONDARY OUTCOMES:
Reactions of folate pathway | 1 year
  Effect of DHFR 19bp deletion on reactions of folate pathway determined in cell culture conditions

CONTACTS AND LOCATIONS:
Overall Officials: Ligi Paul, Ph.D., Principal Investigator — Tufts University

IPD SHARING:
Plan to Share IPD: No